CLINICAL TRIAL: NCT03254459
Title: A Phase 2, Randomized, Open Label, Multiple-Dose, Comparator, Parallel-Group, Safety and Tolerance Study of Buprenorphine Sublingual Spray (0.5 mg TID) Versus Standard of Care Post-Operative Narcotic Therapy for the Treatment of Post-Operative Pain
Brief Title: Study of Buprenorphine Sublingual Spray Versus Standard of Care Narcotic Therapy for the Treatment of Post-Operative Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: INSYS Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INS005-17-111
Record Dates: First submitted 2017-08-16; First posted 2017-08-18 (Actual); Results first posted 2018-10-29 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-09

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Morphine; Oxycodone; Ondansetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Buprenorphine Sublingual Spray 0.5 mg (Experimental): Buprenorphine Sublingual Spray 0.5 milligrams (mg) three times a day (TID) for 7 days.
  Interventions: Drug: Buprenorphine Sublingual Spray; Drug: Zofran
- Standard of Care Narcotic Therapy (Active Comparator): Morphine intravenous (IV), 4 mg TID for 24 hours, followed by oxycodone hydrochloride tablet, 10 mg TID for 6 days.
  Interventions: Drug: Morphine; Drug: Oxycodone Hydrochloride; Drug: Zofran

INTERVENTIONS:
Drug: Buprenorphine Sublingual Spray — 0.5 mg Sublingual Spray
  Arms: Buprenorphine Sublingual Spray 0.5 mg
Drug: Morphine — 4 mg Intravenous Injection
  Arms: Standard of Care Narcotic Therapy
Drug: Oxycodone Hydrochloride — 10 mg tablet
  Arms: Standard of Care Narcotic Therapy
Drug: Zofran — 4 mg oral disintegrating tablet (ODT) or IV injection given at the investigator's discretion for nausea

SUMMARY:
This study will evaluate the safety and tolerability based on the incidence of adverse experiences of buprenorphine sublingual spray (0.5 milligrams [mg] three times daily [TID]) compared with standard post-operative narcotic therapy in participants with postoperative pain. Standard post-operative narcotic therapy is defined as morphine intravenous (IV) injection (4 mg TID) followed by oxycodone hydrochloride tablet (10 mg TID).

ELIGIBILITY:
Inclusion criteria:

1. Is able to speak and understand the language in which the study is being conducted, is able to understand and comply with the procedures and study requirements, and has voluntarily signed and dated an informed consent form approved by an Institutional Review Board before the conduct of any study procedure.
2. Is a male or female ≥18 and ≤65 years of age.
3. Scheduled for elective bunionectomy, breast augmentation (in women only), or abdominoplasty.
4. Is classified using the American Society of Anesthesiologists Physical Status Classification System as P1 to P2.
5. If female, is either not of childbearing potential (defined as postmenopausal for at least 1 year or surgically sterile [bilateral tubal ligation, bilateral oophorectomy, or hysterectomy]) or practicing one of the following medically acceptable methods of birth control:

   1. Hormonal methods such as oral, implantable, injectable, vaginal ring, or transdermal contraceptives for a minimum of 1 full cycle (based on the participant's usual menstrual cycle period) before study drug administration;
   2. Total abstinence from sexual intercourse since the last menses before study drug administration;
   3. Intrauterine device; OR
   4. Double-barrier method (condoms, sponge, or diaphragm with spermicidal jellies or cream).
6. Has a body weight ≥45 kilograms (kg) and a body mass index (BMI) ≤40 kg/m^2.
7. Is willing and able to comply with study requirements (including diet, alcohol, and smoking restrictions), complete evaluations and diary, remain at the study site for ≥72 hours, and return for follow up Day 8 + 2 days after surgery.

Exclusion criteria:

1. Has a known history of allergic reaction or clinically significant intolerance to acetaminophen, aspirin, opioids, or any nonsteroidal anti-inflammatory drugs (NSAIDs); history of NSAID-induced bronchospasm (participants with the triad of asthma, nasal polyps, and chronic rhinitis are at greater risk for bronchospasm and should be considered carefully); or hypersensitivity, allergy, or significant reaction to sulfa (including sulfonamide) medicines, ingredients of the study drug, or any other drugs used in the study, including anesthetics and antibiotics that may be required on the day of surgery.
2. Has experienced any surgical complications or other issues that, in the investigator's opinion, could compromise the participant's safety if he or she continues into randomized treatment or could confound the results of the study.
3. Has a known or suspected history of alcoholism or drug abuse or misuse within 2 years of Screening or evidence of opioid tolerance or physical dependence before dosing with the study drug.
4. Has any clinically significant unstable cardiac, respiratory, neurological, immunological, hematological, or renal disease, or any other condition that, in the investigator's opinion, could compromise the participant's welfare, ability to communicate with the study staff, or otherwise contraindicate study participation.
5. Has long QT Syndrome, a family history of long QT Syndrome, or is taking Class IA or Class III antiarrhythmic medications
6. Has a history or current diagnosis of a significant psychiatric disorder that, in the investigator's opinion, would affect the participant's ability to comply with the study requirements.
7. Has tested positive either on the urine drug screen or on the alcohol Breathalyzer test. Participants who test positive at Screening only and can produce a prescription in their name from their physician for the medication producing the positive test may be considered for study enrollment at the investigator's discretion. However, they must test negative on the day of the surgery.
8. Has a history of a clinically significant (in the investigator's opinion) gastrointestinal (GI) event within 6 months before Screening or has any history of peptic or gastric ulcers or GI bleeding.
9. Has an active infection, mucositis, cold sores, viral lesions, local irritation, or in the investigator's opinion has significant periodontal disease of the oral cavity. In addition, recent (within 1 year) piercing of the tongue or anywhere in the oral cavity.
10. Has a surgical or medical condition of the GI or renal system that, in the investigator's opinion, might significantly alter the absorption, distribution, or excretion of any drug substance.
11. Is considered by the investigator, for any reason (including, but not limited to, the risks described as precautions, warnings, and contraindications in the current version of the investigator's brochure for Buprenorphine Sublingual Spray), to be an unsuitable candidate to receive the study drug.
12. Is receiving systemic chemotherapy, has an active malignancy of any type, or has been diagnosed with cancer within 5 years before Screening (excluding squamous or basal cell carcinoma of the skin).
13. Is currently receiving anticoagulants (eg, heparin or warfarin). Low-dose aspirin for cardioprotection is allowed.
14. Has used drugs known to be a strong inhibitor or inducer of CYP3A4 within 1 week before surgery.
15. Has received a course of systemic corticosteroids (either oral or parenteral) within 1 month before Screening (inhaled nasal steroids and topical corticosteroids are allowed).
16. Has a history of chronic use (defined as daily use for >2 weeks) of NSAIDs, opiates, or glucocorticoids (except inhaled nasal steroids and topical corticosteroids) within 1 month before study drug administration. Aspirin at a daily dose of ≤325 mg is allowed for cardiovascular prophylaxis if the participant has been on a stable dose regimen for ≥30 days before Screening and has not experienced any relevant medical problem.
17. Has a significant renal or hepatic disease, as indicated by clinical laboratory assessment (results ≥3 × the upper limit of normal [ULN] for any liver function test, including aspartate aminotransferase, alanine aminotransferase, and lactate dehydrogenase, or creatinine ≥1.5 × ULN).
18. Has any clinically significant laboratory or 12-lead electrocardiogram finding at Screening that in the investigator's opinion contraindicates study participation.
19. Has screening systolic blood pressure ≥160 mmHg and diastolic blood pressure >100 mmHg (may be repeated one additional time after 5 minutes rest to verify). The investigator may, at his discretion, choose to exclude participants with hypertensive levels lower than these if he deems it in the best interest of the participant.
20. Has a history of sleep apnea or other obstructive airway disease.
21. Has a history of nausea and vomiting with buprenorphine products.
22. Has significant difficulties swallowing capsules or is unable to tolerate oral medication.
23. Previously participated in another clinical study of Buprenorphine Sublingual Spray or received any investigational drug or device or investigational therapy within 30 days before Screening.

Post-surgical eligibility requirements:

The participant will be assessed for the following postoperative eligibility criteria

1. Participants must be awake, breathing spontaneously without significant respiratory depression.
2. Participants must not be actively vomiting or complaining of severe nausea.
3. Participants must be able to answer questions and follow commands.
4. Participants must not have surgical complications that could compromise safety of the participant or confound the results of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2017-11-13 (Actual); Study Completion 2017-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni DeCastro, Study Director — INSYS Therapeutics Inc
Locations (2):
- United States (2):
  - Lotus Clinical Research, LLC, Pasadena, California
  - Epic Medical Research, Murray, Utah

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care Narcotic Therapy: Morphine intravenous (IV), 4 mg TID for 24 hours, followed by oxycodone hydrochloride tablet, 10 mg TID for 6 days.
  Morphine: Morphine
  Oxycodone Hydrochloride: Oxycodone Hydrochloride 10 mg tablet
- Buprenorphine Sublingual Spray 0.5 mg: Buprenorphine Sublingual Spray 0.5 milligrams (mg) three times a day (TID) for 7 days.
  Buprenorphine Sublingual Spray: Buprenorphine Sublingual Spray 0.5 mg
Period: Overall Study
Arm/Group | Standard of Care Narcotic Therapy | Buprenorphine Sublingual Spray 0.5 mg
Started | 50 | 50
Completed | 40 | 27
Not Completed | 10 | 23
Not completed — Adverse Event | 7 | 20
Not completed — Withdrawal by Subject Consent | 3 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Miscellaneous | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care Narcotic Therapy | Buprenorphine Sublingual Spray 0.5 mg | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.2 (10.83) | 37.1 (11.68) | 36.6 (11.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 48 | 96
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 14 | 31
  Not Hispanic or Latino | 33 | 36 | 69
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 3
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 15 | 18 | 33
  White | 29 | 31 | 60
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant administered a pharmaceutical product during the course of a clinical investigation. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of an investigational product, whether or not thought to be related to the investigational product. A TEAE is an AE with onset that occurs after receiving study drug.
Time Frame: Days 1 to 8
Population: Safety population, all participants who received study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Narcotic Therapy | Buprenorphine Sublingual Spray 0.5 mg
Number analyzed (Participants) | 50 | 50
Participants | 33 | 47

2. Secondary Outcome: Percentage of Participants Provided Rescue Medication for Nausea
Description: Zofran was used at the clinician's discretion as rescue medication for nausea.
Time Frame: Days 1 to7
Population: Safety population, all participants who received study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Standard of Care Narcotic Therapy | Buprenorphine Sublingual Spray 0.5 mg
Number analyzed (Participants) | 50 | 50
percentage of participants | 12 | 35

3. Secondary Outcome: Time to First Use of Rescue Medication for Nausea Following Each Dose of the Investigational Product (IP)
Description: Zofran was used at the clinician's discretion as rescue medication for nausea. Time "0" is defined as the time of the administration of study drug.
Time Frame: Days 1 to 7
Population: Safety population, all participants who received study drug.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Standard of Care Narcotic Therapy | Buprenorphine Sublingual Spray 0.5 mg
Number analyzed (Participants) | 50 | 50
hours | NA [NA to NA] — Data could not be calculated as more than 50% of subjects discontinued prior to Day 8. | 11.25 [5.60 to 23.13]

4. Secondary Outcome: Total Use of Rescue Medication for Nausea Over 0 to 24 Hours, Over 0 to 48 Hours, Over 0-72 Hours and 0-7 Days
Description: Zofran was used at the clinician's discretion as rescue medication for nausea. The total use of rescue medication was calculated for the following 4 time-frames: 0 to 24 hours, 0 to 48 hours, 0 to 72 hours and 0 to 7 days.
Time Frame: 0 to 24 hours, 0 to 48 hours, 0 to 72 hours and 0 to 7 days
Population: Safety population, all participants who received study drug.
Measure: Number; unit: cumulative number of rescue doses
Arm/Group | Standard of Care Narcotic Therapy | Buprenorphine Sublingual Spray 0.5 mg
Number analyzed (Participants) | 50 | 50
cumulative number of rescue doses
  0 to 24 hours | 9 | 68
  0 to 48 hours | 18 | 92
  0 to 72 hours | 22 | 110
  0 to 7 days | 42 | 152

5. Secondary Outcome: Pulse Oximetry Levels at 90 Minutes,12, 24, 48 and 72 Hours
Description: Pulse oximetry is a non-invasive method to measure a person's oxygen saturation.
Time Frame: 90 Minutes,12, 24, 48 and 72 Hours
Population: Safety population, all participants who received study drug.
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Arm/Group | Standard of Care Narcotic Therapy | Buprenorphine Sublingual Spray 0.5 mg
Number analyzed (Participants) | 50 | 50
percentage of oxygen saturation
  90 minutes | 96.3 (1.99) | 96.0 (2.11)
  12 hours: number analyzed (Participants) | 50 | 49
  12 hours | 96.0 (1.93) | 95.8 (2.06)
  24 hours: number analyzed (Participants) | 50 | 48
  24 hours | 96.9 (1.63) | 96.6 (2.27)
  48 hours: number analyzed (Participants) | 48 | 46
  48 hours | 96.5 (2.01) | 96.0 (2.15)
  72 hours | 97.3 (1.36) | 96.2 (2.66)

6. Secondary Outcome: Number of Participants With Abnormal Electrocardiograms (ECGs) Findings at 90 Minutes,12, 24, 48 and 72 Hours
Description: A standard 12-lead ECG will be performed after the participant is in the supine (lying face up) position for 5 minutes.
Time Frame: Pre-dose and 90 minutes, 12, 24, 48 and 72 hours after first dose
Population: Safety population, all participants who received study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Narcotic Therapy | Buprenorphine Sublingual Spray 0.5 mg
Number analyzed (Participants) | 50 | 50
Participants
  Pre-dose: number analyzed (Participants) | 49 | 49
  Pre-dose | 26 | 32
  90 minutes: number analyzed (Participants) | 50 | 49
  90 minutes | 33 | 30
  12 hours: number analyzed (Participants) | 50 | 49
  12 hours | 31 | 34
  24 hours: number analyzed (Participants) | 49 | 47
  24 hours | 23 | 29
  48 hours: number analyzed (Participants) | 48 | 45
  48 hours | 18 | 25
  72 hours: number analyzed (Participants) | 42 | 37
  72 hours | 14 | 18

7. Secondary Outcome: Number of Participants With Abnormal Oral Cavity Examinations
Description: Study staff will perform a sublingual (under the tongue) assessment, noting the color of mucosa and whether inflammation is present.
Time Frame: Pre-dose and 90 minutes, 12, 24, 48 and 72 hours after first dose on Days 1 to 4 and End of Study Day 8
Population: Safety population, all participants who received study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Narcotic Therapy | Buprenorphine Sublingual Spray 0.5 mg
Number analyzed (Participants) | 50 | 50
Participants
  Pre-dose | 0 | 0
  90 minutes: number analyzed (Participants) | 49 | 50
  90 minutes | 0 | 0
  12 hours: number analyzed (Participants) | 50 | 49
  12 hours | 0 | 0
  24 hours: number analyzed (Participants) | 50 | 48
  24 hours | 0 | 0
  48 hours: number analyzed (Participants) | 46 | 45
  48 hours | 0 | 1
  72 hours: number analyzed (Participants) | 43 | 37
  72 hours | 0 | 0

ADVERSE EVENTS:
Time Frame: Screening to Day 8
Arm/Group | Standard of Care Narcotic Therapy | Buprenorphine Sublingual Spray 0.5 mg
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 1/50
Other Adverse Events (participants affected / at risk) | 33/50 | 47/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care Narcotic Therapy (N=50) | Buprenorphine Sublingual Spray 0.5 mg (N=50)
Hematoma (General disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care Narcotic Therapy (N=50) | Buprenorphine Sublingual Spray 0.5 mg (N=50)
Nausea (Gastrointestinal disorders) | 17 | 39
Vomiting (Gastrointestinal disorders) | 6 | 26
Constipation (Gastrointestinal disorders) | 4 | 4
Dizziness (Nervous system disorders) | 5 | 11
Headache (Nervous system disorders) | 8 | 9
Somnolence (Nervous system disorders) | 2 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 14
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-08-02): https://cdn.clinicaltrials.gov/large-docs/59/NCT03254459/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-08): https://cdn.clinicaltrials.gov/large-docs/59/NCT03254459/SAP_001.pdf